CLINICAL TRIAL: NCT00015080
Title: Naltrexone in Treatment of Cocaine Dependence
Brief Title: Naltrexone in Treatment of Cocaine Dependence - 5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Cincinnati MDRU (Other)
Purpose: Treatment
Other Study IDs: NIDA-5-0012-5; Y01-5-0012-5
Record Dates: First submitted 2001-04-18; First posted 2001-04-18 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 1996-12

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Naltrexone

INTERVENTIONS:
Drug: Naltrexone

SUMMARY:
The purpose of this study is to determine the efficacy of naltrexone in the treatment of cocaine dependence as measured by: 1) decreased urine benzoylecgonine (BE) levels, 2) decreased cocaine use by self-report, 3) decreased cocaine craving, and 4) retention in treatment.

DETAILED DESCRIPTION:
Double-blind, placebo controlled study of the safety and efficacy of naltrexone in treating cocaine dependence in a patient sample that initiated the study while in an inpatient setting and were then followed-up for 3 months as outpatients.

ELIGIBILITY:
Inclusion Criteria:

1. Meet DSM-III-R criteria for cocaine dependency,
2. 18 to 65 years of age,
3. capable of understanding the study,
4. voluntarily signed consent,
5. male or non-pregnant female using approved form of birth control.

Exclusion Criteria:

1. abnormal liver function tests (SGOT, SGPT, or GGT greater than twice the normal values),
2. opioid use within the last 7 days,
3. use of neuroleptics,
4. having a severe acute medical problem,
5. unable to complete psychiatric rating scales, or
6. judged by the investigator to be unlikely to comply with the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 1995-05; Primary Completion 1996-06 (Actual); Study Completion 1996-07 (Actual)

PRIMARY OUTCOMES:
Retention
Cocaine use
Depression
Anxiety
Addiction severity
Global improvement
Psychopathology

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Somoza, M.D., Ph.D., Principal Investigator — Cincinnati MDRU
Locations (1):
- Cincinnati MDRU, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Somoza, E., et al. A Double-Blind,Placebo Controlled Clinical Trial of Naltrexone as a Treatment for Cocaine Dependence. NIDA Research Monograph, 1998, 179, p. 295.. None